CLINICAL TRIAL: NCT02028117
Title: A Clinical Study Of Enadenotucirev: Dose Finding and Proof of Concept in Platinum-Resistant Epithelial Ovarian Cancer.
Brief Title: Phase I / Dose Expansion Study of Enadenotucirev in Ovarian Cancer Patients
Acronym: OCTAVE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ColoAd1-2001
Record Dates: First submitted 2014-01-03; First posted 2014-01-06 (Estimated); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Recurrent Platinum Resistant Ovarian Cancer
MeSH Terms: interventions — enadenotucirev

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enadenotucirev (Experimental)
  Interventions: Biological: Enadenotucirev

INTERVENTIONS:
Biological: Enadenotucirev — Oncolytic Virus

SUMMARY:
This study is a Phase I / Dose Expansion open label clinical study in patients with platinum-resistant epithelial ovarian cancer. The Phase Ia part of the study will determine the dose of enadenotucirev to be recommended for further studies and will examine primarily the safety and tolerability but also the pharmacokinetics of administering enadenotucirev intraperitoneally. In Phase Ib, the safety and tolerability and the pharmacokinetics of administering enadenotucirev intravenously in combination with weekly paclitaxel will be determined. The Dose Expansion Phase will begin as an open label dose expansion of that regimen and aims to determine whether intravenous enadenotucirev in combination with weekly paclitaxel has a risk benefit profile that supports further investigation in the treatment of patients with platinum-resistant epithelial ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol
2. Age ≥ 18 years
3. Histologically confirmed non-resectable epithelial ovarian, fallopian tube or primary peritoneal cancer
4. Phase Ia and Phase Ib (first 3 patients):

   Confirmed relapsed within the platinum-resistant time frame.
   * Platinum-resistance is defined as progression within 6 months of receiving prior platinum-containing chemotherapy, with progression identified either by CT scanning (RECIST v1.1) or symptomatic CA-125 progression (GCIG CA-125 criteria)
   * The treatment immediately prior to study entry need not be platinum-based OR Absence of other available treatment option

   Phase Ib (after first 3 patients) and Dose Expansion Phase:

   Confirmed relapsed within the platinum-resistant time frame
   * Platinum-resistance is defined as progression within 6 months of receiving prior platinum-containing chemotherapy, with progression identified either by CT scanning (RECIST v1.1) or symptomatic CA-125 progression (GCIG CA-125 criteria)
   * The treatment immediately prior to study entry need not be platinum-based

   Phase Ia and Phase Ib (first 3 patients):

   Evaluable disease (by RECIST v1.1).

   Phase Ib (after first 3 patients) and Dose Expansion Phase:

   Measurable disease (by RECIST v1.1)
5. Able to undergo IP injection, including all administration procedures e.g. placement of IP catheter, iatrogenic ascites and ascites drainage and comply with study procedures in the Investigator's opinion (only required for patients scheduled for IP administration)
6. Recovered to at least grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancy at time of first administration of enadenotucirev
7. ECOG Performance Status Score of 0 - 1
8. Non-impaired renal function

   • Creatinine ≤1.5 mg/dl and estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2 (or measured creatinine clearance ≥60 ml/min)
9. Urine dipstick for proteinuria at screening and baseline negative or trace. Patients may be included with results of 1+ if they have a spot urinary albumin:creatinine ratio (ACR) of either (i) ≤3 mg/mmol or (ii) >3 mg - <70 mg/mmol with a 24 hour urinary protein <0.2 g/24hours Adequate hepatic function

   * Serum bilirubin <1.5 x upper limit of normal (ULN)
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤3 x ULN
10. Adequate bone marrow function:

    * Absolute neutrophil count (ANC) ≥1.5 x 109/l
    * Platelets ≥100 x 109/l
    * Haemoglobin ≥90 g/l
11. Adequate coagulation tests: INR ≤1.5 x ULN;
12. [Criterion has been removed in the current version of the protocol]
13. For females of childbearing potential, a negative pregnancy test must be documented prior to enrolment
14. For women who are not postmenopausal (12 months of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use two adequate methods of contraception, including at least one method with a failure rate of < 1% per year (e.g. hormonal implants, combined oral contraceptives, vasectomised partner), during the treatment period and for at least 3 months after the last dose of study drug
15. For selected patients in the Phase Ia and Dose Expansion Phase part of the study participating in the exploratory assessment of tumour samples:

    • Disease amenable to percutaneous image-guided biopsy.
16. Normal serum complement (C3/C4)

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for enrolment:

1. Tumours of malignant mixed mesodermal (MMMT) or mucinous subtypes, or non-epithelial ovarian cancers (e.g. Brenner tumours, Sex-cord tumours)
2. [Criterion 2 has been removed in the current version of the protocol]
3. Symptomatic sub-acute bowel obstruction, characterised by e.g. regular bloating, nausea, vomiting, constipation or diarrhoea
4. Pregnant or lactating (nursing) women
5. Known and/or a history or evidence of significant immunodeficiency due to underlying illness (e.g. human immunodeficiency virus [HIV]/acquired immunodeficiency syndrome [AIDS]) and/or medication (e.g. systemic corticosteroids at doses higher than dexamethasone 20 mg [or other corticosteroid equivalent to dexamethasone dose] for 14 days or prolonged administration [>14 days] of dexamethasone at doses higher than 10 mg but 20 mg [or other corticosteroid equivalent to dexamethasone dose] or other immunosuppressive medications including cyclosporine, azathioprine, interferons, within the past 14 days)
6. Complete splenectomy
7. Prior allogeneic or autologous bone marrow or organ transplantation
8. Active infections requiring antibiotics, physician monitoring, or recurrent fevers >38.0 degrees centigrade associated with a clinical diagnosis of active infection
9. Active viral disease, positive serology for HIV, hepatitis B or hepatitis C
10. Use of the following anti-viral agents:

    * Ribavirin, adefovir, lamivudine or cidofovir within 7 days prior to day 1
    * or pegylated interferon (PEG-IFN) (within 14 days prior to day 1)
11. Administration of an investigational drug within 28 days
12. Concurrent administration of any cancer therapy other than planned study treatment
13. Major surgery within 2 weeks prior to first dose of enadenotucirev
14. Phase Ib (after first 3 patients) and Dose Expansion Phase only: another primary malignancy within the past 3 years (except for non-melanoma skin cancer or cervical cancer in situ or in situ stage 1 synchronous endometrial cancer)
15. Symptomatic central nervous system (CNS) metastasis
16. Inflammatory diseases of the bowel
17. Concurrent congestive heart failure or prior history of New York Heart Association (NYHA) class III/IV cardiac disease
18. Any condition or illness that, in the opinion of the Investigator or the medical monitor, would compromise patient safety or interfere with the evaluation of the safety of the drug
19. Known allergy to treatment medication or its excipients
20. Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.
21. Any history of renal disease or renal injury or autoimmune disease. Patients with active, known or suspected auto-immune disease or a syndrome that requires systemic or immunosuppressive agents; patients with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune disease only requiring hormone replacement, psoriasis not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger are permitted to enrol providing they comply with the other eligibility criteria relating to renal function)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2019-11-19 (Actual)

PRIMARY OUTCOMES:
Phase I - maximum tolerated dose | Up to day 50 (post first dose)
  The maximally-tolerated dose (MTD) and/or the dose of enadenotucirev recommended for further studies of enadenotucirev when administered as monotherapy by IP injection or as combination therapy by IV infusion with weekly paclitaxel in patients with recurrent, platinum-resistant ovarian cancer.

CONTACTS AND LOCATIONS:
Locations (8):
- Spain (5):
  - Hospital Universitari de Girona Dr. Josep Trueta, Girona
  - Clara Campal Comprehensive Cancer Center Hospital, Madrid
  - MD Anderson Cancer Center, Madrid
  - START MADRID-FJD, Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Miguel Servet, Zaragoza
- United Kingdom (3):
  - The Royal Surrey County Hospital, Guildford, Surrey
  - Beatson Institute, Glasgow
  - The Christie Hospital, Manchester

REFERENCES:
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458
- [Derived] Moreno V, Barretina-Ginesta MP, Garcia-Donas J, Jayson GC, Roxburgh P, Vazquez RM, Michael A, Anton-Torres A, Brown R, Krige D, Champion B, McNeish I. Safety and efficacy of the tumor-selective adenovirus enadenotucirev with or without paclitaxel in platinum-resistant ovarian cancer: a phase 1 clinical trial. J Immunother Cancer. 2021 Dec;9(12):e003645. doi: 10.1136/jitc-2021-003645. PMID 34893524
- See also: OCTAVE results as listed on EudraCT — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-001276-38/results